CLINICAL TRIAL: NCT06172101
Title: Prospective Evaluation of Improvement in Pain and Quality of Life After Free Fat Flap for Treatment of Recurrent Neurological Thoracobrachial Outlet Syndrome
Brief Title: Free Fat Flap In Recurrent Neurogenic Thoracic Outlet Syndrome Surgical Treatment
Acronym: FIRST
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_UL_001
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Neurogenic Thoracic Outlet Syndrome
Keywords: Recurrent neurogenic thoracic outlet syndrome; Free fat flap
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Free fat flap — Free fat flap In Recurrent neurogenic thoracic outlet syndrome Surgical Treatment

SUMMARY:
The Thoraco-Brachial Outlet Syndrome (T-BOS) corresponds to the entirety of clinical manifestations related to the compression of the branches of the brachial plexus and/or the subclavian vessels during their passage through the cervico-thoracic region.

Following surgery, a recurrence of symptoms occurs in 5% to 30% of operated patients. The treatment of these recurrences primarily relies on conservative therapies, and in case of failure, surgical intervention, particularly neurolysis of the brachial plexus.

In order to prevent a new recurrence, it is desirable to cover the neurolyzed brachial plexus with a flap, providing better local vascularization. However, fatty perforating flaps, by avoiding muscle harvesting, reduce donor site sequelae. We aim to investigate, through validated and recommended questionnaires, the impact of covering the neurolyzed brachial plexus with a free fatty flap after neurolysis in the context of recurrent neurological Thoraco-Brachial Outlet Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent brachial plexus neurolysis and free fat flap coverage in the context of recurrence of neurological thoraco-brachial outlet syndrome

Exclusion Criteria:

* Patients were unable to express their non-opposition to participating in the study.
* patients under guardianship or trusteeship.
* patients whose mother tongue is not French.
* patients who cannot read and/or write.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients operated on for brachial plexus neurolysis and free fat flap coverage in the setting of recurrent neurological thoracic brachial outlet syndrome.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Evaluating the impact on pain of covering the brachial plexus with a free fat flap | pre-op and six months post-op
  the percentage reduction in pain assessed by a numerical scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Lancien, Nantes, France